CLINICAL TRIAL: NCT03460756
Title: A Phase 2, Double-blind, Placebo-controlled, Multicenter Study to Evaluate Safety, Tolerability, and Efficacy of Oral Administration of Ganaxolone in Women With Postpartum Depression
Brief Title: A Clinical Trial of Oral Ganaxolone in Women With Postpartum Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-PPD-2003
Record Dates: First submitted 2018-01-18; First posted 2018-03-09 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Depressive Disorder; Depression; Depression, Postpartum; Behavioral Symptoms; Mood Disorders; Mental Disorder; Pregnancy Complications; Postpartum Blues; PPD; Postpartum Disorder
Keywords: Postpartum Care; Postpartum Depression
MeSH Terms: conditions — Depressive Disorder; Depression; Depression, Postpartum; Behavioral Symptoms; Mood Disorders; Mental Disorders; Pregnancy Complications; Puerperal Disorders | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ganaxolone (Experimental): Oral
  Interventions: Drug: Ganaxolone
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ganaxolone — Oral
  Arms: Ganaxolone
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
A clinical study to evaluate safety, tolerability and efficacy of oral administration of ganaxolone in women with postpartum depression

ELIGIBILITY:
Inclusion Criteria:

* Experiencing a major depressive episode, which started between the start of the third trimester and 4 weeks following delivery. The major depressive episode must be diagnosed according to Mini International Neuropsychiatric Interview (MINI) 7.0 interview
* Given birth in the last 6 months
* HAMD17 score of ≥ 20 at screening but < 26
* Must agree to stop breastfeeding from start of study treatment or must agree to temporarily cease giving breast milk to her infant(s)

Exclusion Criteria:

* Current history of any psychotic illness, including major depressive episode with psychotic features
* History of suicide attempt within the past 3 years
* History of bipolar I disorder
* History of seizure discorder

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with postpartum depression
Enrollment: 84 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hulihan, MD, Study Director — Marinus Pharmaceuticals
Locations (32):
- United States (32):
  - Marinus Research Site, Glendale, California
  - Marinus Research Site, Lemon Grove, California
  - Marinus Research Site, Long Beach, California
  - Marinus Research Site, Oceanside, California
  - Marinus Research Site, Panorama City, California
  - Marinus Research Site, San Bernardino, California
  - Marinus Research Site, San Marcos, California
  - Marinus Research Site, Ventura, California
  - Marinus Research Site, Gainesville, Florida
  - Marinus Research Site, Hollywood, Florida
  - Marinus Research Site, Jacksonville, Florida
  - Marinus Research Site, North Miami, Florida
  - Marinus Research Site, Atlanta, Georgia
  - Marinus Research Site, Decatur, Georgia
  - Marinus Research Site, Marietta, Georgia
  - Marinus Research Site, Idaho Falls, Idaho
  - Marinus Research Site, Hoffman Estates, Illinois
  - Marinus Research Site, Leawood, Kansas
  - Marinus Research Site, Wichita, Kansas
  - Marinus Research Site, Flowood, Mississippi
  - Marinus Research Site, Las Vegas, Nevada
  - Marinus Research Site, Albuquerque, New Mexico
  - Marinus Research Site, Raleigh, North Carolina
  - Marinus Research Site, Englewood, Ohio
  - Marinus Research Site, Downingtown, Pennsylvania
  - Marinus Research Site, Media, Pennsylvania
  - Marinus Research Site, Houston, Texas
  - Marinus Research Site, Irving, Texas
  - Marinus Research Site, League City, Texas
  - Marinus Research Site, San Antonio, Texas
  - Marinus Research Site, Orem, Utah
  - Marinus Research Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- TID (2-week): Oral ganaxolone doses were titrated over 6 days to a daily dose of 900 milligrams/ day (mg/day) (3 divided doses) and was maintained until Day 10, followed by a taper over 4 days
- QHS (2-week): Oral ganaxolone doses were titrated to a daily dose of 675 mg/day approximately 10 PM or before going to bed for the night (QHS) over 4 days, which was maintained until Day 10, followed by a taper over 4 days
- QHS (4-week): Oral ganaxolone doses were titrated to a daily dose of 675 mg/day QHS for 28 days, followed by a taper over 4 days.
- 1125 mg (4-week): Oral ganaxolone was dosed as 675 mg at approximately 7 PM or with supper (Q7PM) and QHS (for a total of 1,350 mg/day on the first 2 days), followed by a daily dose of 1,125 mg/day at Q7PM for 26 days and a taper over 4 days
Period: Overall Study
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Started | 2 | 14 | 25 | 43
Completed (2-week TID group was discontinued after 2 subjects were enrolled due to daytime TEAE of sedation and dizziness) | 2 | 9 | 16 | 34
Not Completed | 0 | 5 | 9 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 7 | 3

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- TID (2-week): Oral ganaxolone doses were titrated to a daily dose of 900 mg/day Oral ganaxolone doses were titrated to a daily dose of 675 mg/day QHS over 4 days, which was maintained until Day 10, followed by a taper over 4 days
- QHS (2-week): Oral ganaxolone doses were titrated to a daily dose of 675 mg/day QHS over 4 days, which was maintained until Day 10, followed by a taper over 4 days
- QHS (4-week): Oral ganaxolone was dosed at a daily dose of 675 mg/day QHS for 28 days, followed by a taper over 4 days
- Total: Total of all reporting groups
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week) | Total
Number analyzed (Participants) | 2 | 14 | 25 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (7.78) | 27.5 (7.27) | 27.4 (5.27) | 28.0 (5.72) | 27.7 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 14 | 25 | 43 | 84
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 11 | 12 | 27
  Not Hispanic or Latino | 1 | 11 | 14 | 31 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 4 | 10 | 16 | 31
  White | 1 | 7 | 13 | 25 | 46
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale 17-item Version (HAMD17) Through Treatment
Description: The HAMD17 was a 17-item clinician-rated instrument used to assess the range of symptoms that were most frequently observed in participants with major depression. All items were scored on an ordinal scale between 0 and 4 (8 items) or 0 and 2 (9 items) of increasing severity. Each of 17 items was rated by clinician with rating of 0: absent, 1: doubtful to mild, 2: mild to moderate, 3: moderate to severe, and 4: very severe. A total score (0 to 52) was calculated by adding scores of all 17 items, where 0 indicated no depression and 52 indicated severe depression. Higher score represented more severe condition. Baseline was defined as the Day 1 assessment before study drug infusion. Change from Baseline is defined as post dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and through Day 10 for 2 week treatment group and Day 29 for 4 week treatment groups
Population: Safety Set was defined as all participants who were dispensed study drug. Only those participants with HAMD17 response through treatment have been presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- TID (2-week): Oral ganaxolone doses were titrated to a daily dose of 900 mg/day (in 3 divided doses) and was maintained until Day 10, followed by a taper over 4 days
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Number analyzed (Participants) | 2 | 13 | 23 | 42
score on a scale
  Day 2/4: number analyzed (Participants) | 2 | 13 | 22 | 42
  Day 2/4 | -8.0 (9.90) | -5.7 (4.87) | -0.8 (3.19) | -2.6 (5.46)
  Day 7: number analyzed (Participants) | 2 | 10 | 0 | 0
  Day 7 | -15.0 (12.73) | -6.7 (7.93) |  |
  Day 8/10: number analyzed (Participants) | 1 | 10 | 23 | 39
  Day 8/10 | -3.0 (0) | -10.5 (7.21) | -6.8 (7.25) | -10.2 (7.44)
  Day 15/17: number analyzed (Participants) | 2 | 11 | 21 | 39
  Day 15/17 | -9.5 (9.19) | -8.8 (7.12) | -9.7 (7.36) | -9.4 (7.94)
  Day 22: number analyzed (Participants) | 0 | 0 | 19 | 37
  Day 22 |  |  | -10.3 (5.94) | -12.0 (7.98)
  Day 29: number analyzed (Participants) | 0 | 0 | 21 | 35
  Day 29 |  |  | -12.2 (8.40) | -14.0 (7.64)

2. Secondary Outcome: Change From Baseline in Hamilton Depression Rating Scale 17-item Version Post Treatment
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Through Day 38 for 2 week treatment group and Day 71 and 119 for 4 week treatment groups
Population: Safety Set. Only those participants with HAMD17 response post treatment have been presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Number analyzed (Participants) | 2 | 8 | 20 | 36
score on a scale
  Day 36/38 | -19.0 (7.07) | -7.1 (8.44) | -14.6 (9.63) | -12.4 (8.82)
  Day 57/59: number analyzed (Participants) | 0 | 0 | 17 | 36
  Day 57/59 |  |  | -13.2 (8.20) | -12.3 (9.11)
  Day 71: number analyzed (Participants) | 0 | 0 | 0 | 31
  Day 71 |  |  |  | -12.2 (8.45)
  Day 89: number analyzed (Participants) | 0 | 0 | 18 | 0
  Day 89 |  |  | -14.2 (9.98) |
  Day 119: number analyzed (Participants) | 0 | 0 | 11 | 0
  Day 119 |  |  | -20.5 (6.59) |

3. Secondary Outcome: Number of Participants With Response to Hamilton Depression Rating Scale 17 Item (HAMD17)
Description: HAMD17 Response was defined as ≥50% reduction from Baseline in total score. The HAMD-17 is a 17-item assessment used to assess the severity of depression and its improvement during the course of therapy. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Items rated on the 3-point scale include: insomnia early, middle, late; somatic symptoms gastrointestinal and general; genital symptoms; loss of weight; insight. Items rated on 5-point scale include: depressed mood; feelings of guilt; suicide; work and activities; retardation; agitation; anxiety psychic and somatic; hypochondriasis. The total score was the sum of the scores from HAMD-17 Items 1 through 17 and ranged from 0 (not at all depressed) to 52 (severely depressed). Higher scores indicate greater symptom severity. Number of participants with response to HAMD-17 has been presented.
Time Frame: Day 2 (all treatment groups), Day 7 (TID & QHS), Day 8/10 (all treatment groups), Day 15/17 (all treatment groups), Day 22 and 29 (QHS, 1125mg), Day 36/38 (all treatment groups), Day 57/59 (QHS, 1125mg), Day 71 (1125mg), Day 89 (QHS), Day 119 (QHS)
Population: Safety Set. Only those participants with data available at specified timepoints have been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Number analyzed (Participants) | 2 | 13 | 23 | 42
Participants
  Day 2/4 - Response: number analyzed (Participants) | 2 | 13 | 22 | 42
  Day 2/4 - Response | 0 | 2 | 0 | 3
  Day 7 - Response: number analyzed (Participants) | 2 | 10 | 0 | 0
  Day 7 - Response | 1 | 4 |  |
  Day 8/10 - Response: number analyzed (Participants) | 1 | 10 | 23 | 39
  Day 8/10 - Response | 0 | 4 | 7 | 12
  Day 15/17 - Response: number analyzed (Participants) | 2 | 11 | 21 | 39
  Day 15/17 - Response | 1 | 4 | 7 | 16
  Day 22 - Response: number analyzed (Participants) | 0 | 0 | 19 | 37
  Day 22 - Response |  |  | 8 | 20
  Day 29 - Response: number analyzed (Participants) | 0 | 0 | 21 | 35
  Day 29 - Response |  |  | 10 | 22
  Day 36/38 - Response: number analyzed (Participants) | 2 | 8 | 20 | 36
  Day 36/38 - Response | 2 | 3 | 12 | 17
  Day 57/59 - Response: number analyzed (Participants) | 0 | 0 | 17 | 36
  Day 57/59 - Response |  |  | 8 | 18
  Day 71 - Response: number analyzed (Participants) | 0 | 0 | 0 | 31
  Day 71 - Response |  |  |  | 13
  Day 89 - Response: number analyzed (Participants) | 0 | 0 | 18 | 0
  Day 89 - Response |  |  | 9 |
  Day 119 - Response: number analyzed (Participants) | 0 | 0 | 11 | 0
  Day 119 - Response |  |  | 10 |

4. Secondary Outcome: Number of Participants With Hamilton Depression Rating Scale 17-item Remission
Description: Remission was defined as an observed total score of 0 to 7. The HAMD-17 is a 17-item assessment used to assess the severity of depression and its improvement during the course of therapy. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Items rated on the 3-point scale include: insomnia early, middle, late; somatic symptoms gastrointestinal and general; genital symptoms; loss of weight; insight. Items rated on 5-point scale include: depressed mood; feelings of guilt; suicide; work and activities; retardation; agitation; anxiety psychic and somatic; hypochondriasis. The total score was the sum of the scores from HAMD-17 Items 1 through 17 and ranged from 0 (not at all depressed) to 52 (severely depressed). Higher scores indicate greater symptom severity. Number of participants with HAMD-17 remission has been presented.
Time Frame: Day 8/10 (all treatment arms), Day 15/17 (all treatment arms), Day 22 and 29 (QHS & 1125mg), Day 36/38 (all treatment arms), Day 57/59 (QHS & 1125mg), Day 71 (1125mg), Day 89 & 119 (QHS)
Population: Safety Set. Only those participants with data available at specified timepoints have been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Number analyzed (Participants) | 2 | 11 | 23 | 39
Participants
  Day 8/10 - Remission: number analyzed (Participants) | 1 | 10 | 23 | 39
  Day 8/10 - Remission | 0 | 1 | 1 | 8
  Day 15/17 - Remission: number analyzed (Participants) | 2 | 11 | 21 | 39
  Day 15/17 - Remission | 0 | 2 | 4 | 8
  Day 22 - Remission: number analyzed (Participants) | 0 | 0 | 19 | 37
  Day 22 - Remission |  |  | 3 | 10
  Day 29 - Remission: number analyzed (Participants) | 0 | 0 | 21 | 35
  Day 29 - Remission |  |  | 7 | 14
  Day 36/38 - Remission: number analyzed (Participants) | 2 | 8 | 20 | 36
  Day 36/38 - Remission | 1 | 1 | 9 | 11
  Day 57/59 - Remission: number analyzed (Participants) | 0 | 0 | 17 | 36
  Day 57/59 - Remission |  |  | 5 | 12
  Day 71 - Remission: number analyzed (Participants) | 0 | 0 | 0 | 31
  Day 71 - Remission |  |  |  | 9
  Day 89 - Remission: number analyzed (Participants) | 0 | 0 | 18 | 0
  Day 89 - Remission |  |  | 7 |
  Day 119 - Remission: number analyzed (Participants) | 0 | 0 | 11 | 0
  Day 119 - Remission |  |  | 8 |

5. Secondary Outcome: Change From Baseline in Edinburgh Postnatal Depression Scale (EPDS) Total Score
Description: The EPDS is a validated 10-question depression assessment for postpartum women, which includes anxiety symptoms and excludes constitutional symptoms associated with depression common in the postpartum period, such as changes in sleeping patterns. It consists of 10 multiple choice questions with scores for each question ranging from 0-3. Questions 1, 2, & 4 are scored 0, 1, 2 or 3 with top box scored as 0 and the bottom box scored as 3. Questions 3 and 5 to 10 are reverse scored, with the top box scored as a 3 and the bottom box scored as 0. Scores are then summed for a total score, which ranges from 0: no depression to 30: severe depression. Higher score indicates severe depression. Baseline was defined as the Day 1 assessment before study drug infusion. Change from Baseline is defined as post dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) through Day 119
Population: Safety Set. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Number analyzed (Participants) | 2 | 12 | 24 | 42
Score on a scale
  Day 2/4: number analyzed (Participants) | 2 | 12 | 22 | 42
  Day 2/4 | -0.5 (2.12) | -1.4 (2.19) | -0.8 (1.18) | -0.6 (1.64)
  Day 7: number analyzed (Participants) | 2 | 10 | 0 | 0
  Day 7 | -2.0 (2.83) | -2.3 (2.06) |  |
  Day 8/10: number analyzed (Participants) | 1 | 10 | 24 | 39
  Day 8/10 | -3.0 (NA) — NA indicates standard error could not be calculated for single participant. | -1.3 (1.57) | -1.5 (1.74) | -2.3 (2.01)
  Day 15/17: number analyzed (Participants) | 2 | 11 | 20 | 40
  Day 15/17 | -5.0 (0.00) | -2.6 (1.63) | -1.8 (2.17) | -2.2 (2.38)
  Day 22: number analyzed (Participants) | 0 | 0 | 20 | 36
  Day 22 |  |  | -2.7 (2.18) | -3.0 (2.62)
  Day 29: number analyzed (Participants) | 0 | 0 | 21 | 38
  Day 29 |  |  | -2.9 (2.79) | -3.1 (2.77)
  Day 36/38: number analyzed (Participants) | 2 | 8 | 20 | 36
  Day 36/38 | -2.0 (2.83) | -2.6 (1.85) | -3.1 (2.77) | -3.7 (2.64)
  Day 57/59: number analyzed (Participants) | 0 | 0 | 19 | 36
  Day 57/59 |  |  | -2.5 (2.46) | -3.4 (2.68)
  Day 71: number analyzed (Participants) | 0 | 0 | 0 | 32
  Day 71 |  |  |  | -3.3 (2.31)
  Day 89: number analyzed (Participants) | 0 | 0 | 19 | 0
  Day 89 |  |  | -2.6 (2.41) |
  Day 119: number analyzed (Participants) | 0 | 0 | 14 | 0
  Day 119 |  |  | -3.3 (3.20) |

6. Secondary Outcome: Change From Baseline in Spielberger State-Trait Anxiety Inventory, 6-item Version
Description: The Spielberger State-Trait Anxiety Inventory was a 6-item questionnaire designed and validated. It is a reliable and sensitive measure of anxiety. The 6-item version has been shown to have acceptable reliability, producing similar scores as the full 20-item inventory for those with normal and raised levels of anxiety. Participants are prompted to respond to indicate "how [the participant] feel right now, at this moment", followed by a list of common experiences like "I feel calm, I am tense, I feel upset, I am relaxed I feel content and I am worried." Responses range from Not at all (1) to Very much (4), with overall scores ranging from 20-80, where higher scores reflected higher states of anxiety. Baseline was defined as the Day 1 assessment before study drug infusion. Change from Baseline is defined as post dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) through Day 119
Population: Safety Set. Only those participants with data available at specified timepoints has been analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Number analyzed (Participants) | 2 | 12 | 24 | 42
Scores on a scale
  Day 2/4: number analyzed (Participants) | 2 | 12 | 22 | 42
  Day 2/4 | -11.7 (11.81) | -6.4 (11.77) | -1.8 (11.45) | -9.9 (14.84)
  Day 7: number analyzed (Participants) | 2 | 10 | 0 | 0
  Day 7 | -11.7 (7.00) | -9.0 (11.86) |  |
  Day 8/10: number analyzed (Participants) | 1 | 10 | 24 | 39
  Day 8/10 | -20.0 (NA) — NA indicates standard error could not be calculated for single participant. | -5.7 (11.00) | -11.8 (12.40) | -16.8 (17.53)
  Day 15/17: number analyzed (Participants) | 2 | 11 | 20 | 40
  Day 15/17 | -33.3 (9.48) | -14.8 (13.45) | -14.5 (17.58) | -15.2 (19.97)
  Day 22: number analyzed (Participants) | 0 | 0 | 20 | 36
  Day 22 |  |  | -13.0 (17.48) | -21.8 (19.81)
  Day 29: number analyzed (Participants) | 0 | 0 | 21 | 38
  Day 29 |  |  | -17.13 (17.94) | -21.4 (20.34)
  Day 36/38: number analyzed (Participants) | 2 | 8 | 20 | 36
  Day 36/38 | -31.7 (2.33) | -11.3 (5.31) | -20.5 (17.62) | -23.2 (18.96)
  Day 57/59: number analyzed (Participants) | 0 | 0 | 19 | 36
  Day 57/59 |  |  | -16.3 (15.52) | -22.8 (19.72)
  Day 71: number analyzed (Participants) | 0 | 0 | 0 | 32
  Day 71 |  |  |  | -19.2 (18.75)
  Day 89: number analyzed (Participants) | 0 | 0 | 19 | 0
  Day 89 |  |  | -14.7 (18.52) |
  Day 119: number analyzed (Participants) | 0 | 0 | 14 | 0
  Day 119 |  |  | -16.7 (17.45) |

7. Secondary Outcome: Number of Participants With Clinical Global Impression-Improvement
Description: The CGI-I scale is a clinician-rated 7-point scale used to assess how much the participant's illness had improved or worsened relative to a Baseline state at the beginning of the intervention. It was rated as: 1. "very much improved" 2. "much improved" 3. "minimally improved" 4. "no change" 5. "minimally worse" 6. "much worse" 7. "very much worse". Higher scores indicated worse condition. Only those participants with CGI- improvement have been presented.
Time Frame: Baseline through Day 119
Population: Safety Set. Only those participants with data available at specified timepoints has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
Number analyzed (Participants) | 2 | 14 | 25 | 43
Participants
  Day 2/4 - Very much Improved: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 2/4 - Much Improved: number analyzed (Participants) | 2 | 13 | 22 | 42
  Day 2/4 - Much Improved | 0 | 1 | 1 | 4
  Day 2/4 - Minimally Improved: number analyzed (Participants) | 2 | 13 | 22 | 42
  Day 2/4 - Minimally Improved | 1 | 6 | 4 | 15
  Day 7 - Very much Improved: number analyzed (Participants) | 2 | 10 | 0 | 0
  Day 7 - Very much Improved | 0 | 1 |  |
  Day 7 - Much Improved: number analyzed (Participants) | 2 | 10 | 0 | 0
  Day 7 - Much Improved | 1 | 5 |  |
  Day 7 - Minimally Improved: number analyzed (Participants) | 2 | 10 | 0 | 0
  Day 7 - Minimally Improved | 1 | 2 |  |
  Day 8/10 - Very much Improved: number analyzed (Participants) | 1 | 10 | 0 | 39
  Day 8/10 - Very much Improved | 0 | 2 |  | 3
  Day 8/10 - Much Improved: number analyzed (Participants) | 1 | 10 | 24 | 39
  Day 8/10 - Much Improved | 1 | 5 | 7 | 14
  Day 8/10 - Minimally Improved: number analyzed (Participants) | 1 | 10 | 24 | 39
  Day 8/10 - Minimally Improved | 0 | 2 | 8 | 11
  Day 15/17 - Very much Improved: number analyzed (Participants) | 2 | 11 | 20 | 40
  Day 15/17 - Very much Improved | 0 | 2 | 1 | 6
  Day 15/17 - Much Improved: number analyzed (Participants) | 2 | 11 | 20 | 40
  Day 15/17 - Much Improved | 2 | 5 | 9 | 15
  Day 15/17 - Minimally Improved: number analyzed (Participants) | 2 | 11 | 20 | 40
  Day 15/17 - Minimally Improved | 0 | 3 | 5 | 9
  Day 22 - Very much Improved: number analyzed (Participants) | 0 | 0 | 20 | 37
  Day 22 - Very much Improved |  |  | 1 | 7
  Day 22 - Much Improved: number analyzed (Participants) | 0 | 0 | 20 | 37
  Day 22 - Much Improved |  |  | 9 | 16
  Day 22 - Minimally Improved: number analyzed (Participants) | 0 | 0 | 20 | 37
  Day 22 - Minimally Improved |  |  | 6 | 6
  Day 29 - Very much Improved: number analyzed (Participants) | 0 | 0 | 21 | 37
  Day 29 - Very much Improved |  |  | 4 | 11
  Day 29 - Much Improved: number analyzed (Participants) | 0 | 0 | 21 | 37
  Day 29 - Much Improved |  |  | 7 | 16
  Day 29 - Minimally Improved: number analyzed (Participants) | 0 | 0 | 21 | 37
  Day 29 - Minimally Improved |  |  | 8 | 5
  Day 36/38 - Very much Improved | 0 | 1 | 8 | 12
  Day 36/38 - Much Improved | 2 | 3 | 4 | 10
  Day 36/38 - Minimally Improved | 0 | 1 | 7 | 10
  Day 57/59 - Very Much Improved: number analyzed (Participants) | 0 | 0 | 19 | 36
  Day 57/59 - Very Much Improved |  |  | 4 | 9
  Day 57/59 - Much Improved: number analyzed (Participants) | 0 | 0 | 19 | 36
  Day 57/59 - Much Improved |  |  | 9 | 14
  Day 57/59 - Minimally Improved: number analyzed (Participants) | 0 | 0 | 19 | 36
  Day 57/59 - Minimally Improved |  |  | 2 | 7
  Day 71 - Very Much Improved: number analyzed (Participants) | 0 | 0 | 0 | 32
  Day 71 - Very Much Improved |  |  |  | 8
  Day 71 - Much Improved: number analyzed (Participants) | 0 | 0 | 0 | 32
  Day 71 - Much Improved |  |  |  | 14
  Day 71 - Minimally Improved: number analyzed (Participants) | 0 | 0 | 0 | 32
  Day 71 - Minimally Improved |  |  |  | 6
  Day 89 - Very much Improved: number analyzed (Participants) | 0 | 0 | 19 | 0
  Day 89 - Very much Improved |  |  | 6 |
  Day 89 - Much Improved: number analyzed (Participants) | 0 | 0 | 19 | 0
  Day 89 - Much Improved |  |  | 4 |
  Day 89 - Minimally Improved: number analyzed (Participants) | 0 | 0 | 19 | 0
  Day 89 - Minimally Improved |  |  | 6 |
  Day 119 - Very Much Improved: number analyzed (Participants) | 0 | 0 | 25 | 0
  Day 119 - Very Much Improved |  |  | 5 |
  Day 119 - Much Improved: number analyzed (Participants) | 0 | 0 | 25 | 0
  Day 119 - Much Improved |  |  | 3 |
  Day 119 - Minimally Improved: number analyzed (Participants) | 0 | 0 | 25 | 0
  Day 119 - Minimally Improved |  |  | 3 |

ADVERSE EVENTS:
Time Frame: Baseline up through Day 119
Arm/Group | TID (2-week) | QHS (2-week) | QHS (4-week) | 1125 mg (4-week)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/14 | 0/25 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/14 | 0/25 | 1/43
Other Adverse Events (participants affected / at risk) | 2/2 | 5/14 | 16/25 | 32/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TID (2-week) (N=2) | QHS (2-week) (N=14) | QHS (4-week) (N=25) | 1125 mg (4-week) (N=43)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TID (2-week) (N=2) | QHS (2-week) (N=14) | QHS (4-week) (N=25) | 1125 mg (4-week) (N=43)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 7
Headache (Nervous system disorders) | 1 | 1 | 4 | 11
Sedation (Nervous system disorders) | 2 | 2 | 3 | 7
Somnolence (Nervous system disorders) | 0 | 0 | 4 | 9
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT03460756/Prot_002.pdf
  • Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT03460756/SAP_003.pdf